CLINICAL TRIAL: NCT03521011
Title: The Role Of Unenhanced MSCT Abdomen in Diagnosis of Causes of Acute Abdomen
Brief Title: Non Enhanced MSCT In Diagnosis of Causes of Acute Abdomen Cases
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Engy Zarief, The Role Of Unenhanced MSCT Abdomen in diagnosis of causes of Acute Abdomen., Assiut University
Other Study IDs: MSCT in Acute Abdomen
Record Dates: First submitted 2018-04-25; First posted 2018-05-11 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Non Enhanced MSCT Abdomen in Diagnosis of Acute Abdomen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MSCT — Non enhanced MSCT Abdomen

SUMMARY:
The acute abdomen is one of the most frequent causes for presentation to the emergency department. Imaging plays an important role for an accurate diagnosis, which in turn diminishes morbidity and mortality Jastaniah and Salih demonstrate optimum CT aspects and emphasize on the important features of CT for those patients presenting with an acute abdominal pain at the Emergency Department. The reported data by this study are based on the author working experience, which forms a continuous protocol adjustment process. The present study provides evidence that CT would result in definite diagnosis of patients with abdominal pain in terms of the detection of some urgent conditions . The acute abdomen may be defined generally as an intra-abdominal process causing severe pain and often requiring medical or surgical intervention. The acute abdomen is a frequent entity at the Emergency Department, the acute abdomen may be life threatening and so rapid diagnosis of patients presenting with acute abdominal pain is required . Diagnostic work-up with imaging can consist of plain X-ray, ultrasonography (US), computed tomography (CT) and even diagnostic laparoscopy. During the last decade, a trend towards increased use of computed tomography in patients with abdominal pain can be seen. In general, acute abdominal pain is responsible for about 10% of total number of patients visiting the emergency. Quick and precise diagnosis for the urgent cases is usually vital for treatment. Medical imaging is commonly used for the diagnosis of most acute abdomen pain. Abdomen and pelvis are reviewed by CT scan. Specifically, in cases of acute abdomen complain.

DETAILED DESCRIPTION:
There is no gold standard for diagnosis of acute abdomen as it still a matter of cooperation between clinical data, radiological and laboratory worker. The aim of this study was to demonstrate optimum CT aspects and emphasize on the important features of CT for those patients presenting with an acute abdominal pain clinically suspected to have emergency operation .

ELIGIBILITY:
Inclusion Criteria:

* Any Case Of Acute Abdominal Pain suspected to be surgical cases in adults.

Exclusion Criteria:

* If pediatric .
* If associated with pregnancy.
* The patient have severe cardiac or respiratory disease ,cant to lie supine.
* If suspected medical case of acute abdomen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of this study is to improve diagnostic efficiency dealing with acute abdomen not to stabilize a new technique.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis causes of Acute Abdomen By using Non enhanced MSCT Abdomen | baseline
  Diagnosis causes of Acute Abdomen By using Non enhanced MSCT Abdomen and compare with operative data and laboratory result.

CONTACTS AND LOCATIONS:
Locations (1):
- Engy zarief Zarief, Asyut, Resident Doctor, Egypt